CLINICAL TRIAL: NCT02568735
Title: The Central Nervous Penetration of Dexketoprofen and Etoricoxib and Their Effect on Pain and Inflammatory Reaction in Patients Undergoing Hip Arthroplasty
Brief Title: Dexketoprofen and Etoricoxib in Patients Undergoing Hip Arthroplasty
Acronym: etoketo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH30062008
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Pain, Postoperative
Keywords: Dexketoprofen; Etoricoxib; hip arthroplasty; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — dexketoprofen trometamol; Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etoricoxib (Experimental): Etoricoxib 60mg if body weight≤ 60kg, 90mg if body weight 61-90kg and 120mg if body weight> 90kg by mouth
  Interventions: Drug: Etoricoxib
- Dexketoprofen (Active Comparator): Dexketoprofen 0,5 mg/kg up to 50 mg intravenously
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Dexketoprofen — After total hip replacement surgery patient were given either etoricoxib or dexketoprofen
  Arms: Dexketoprofen
Drug: Etoricoxib — After total hip replacement surgery patient were given either etoricoxib or dexketoprofen
  Arms: Etoricoxib

SUMMARY:
The main purpose of this study was to determine the plasma and central nervious system pharmacokinetics of dexketoprofen and etoricoxib. The secondary aim was to asses their effect on the concentrations of interleukin 6, prostaglandin E2 and other proinflammatory markers both in plasma and cerebrospinal fluid. Thirdly, the investigators aimed to evaluate their efficacy in postoperative pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* agreed to participate the study
* American Society of Anesthesiologist s physical status classification 1-3
* elective hip arthroplasty planned
* no contraindications to the study drugs
* no contraindication to lumbar puncture

Exclusion Criteria:

* refused to participate the study
* age less than 40 or over 75 years
* Planned anesthesia method other than spinal anesthesia
* contraindications to the study drugs
* Contraindications to lumbar puncture

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid concentration dexketoprofen and etoricoxib | 0-24 hours
  Cerebrospinal fluid concentration of dexketoprofen and etoricoxib
Plasma concentration dexketoprofen and etoricoxib | 0-24 hours
  Plasma concentration dexketoprofen and etoricoxib

SECONDARY OUTCOMES:
Pain | 0-24 h
  Pain assessed with numeral rating scale

IPD SHARING:
Plan to Share IPD: No